CLINICAL TRIAL: NCT04802889
Title: Microarchitecture of Vitreoretinal Contact
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The S.N. Fyodorov Eye Microsurgery State Institution (Other Government)
Responsible Party: Principal Investigator, Lyskin Pavel Vladimirovich, MD, PhD, MD, PhD, ophthalmosurgeon, The S.N. Fyodorov Eye Microsurgery State Institution
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 124576
Record Dates: First submitted 2020-12-06; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Vitreoretinal Detachment; Vitreo-Retinal Adhesion
Keywords: internal limiting membrane; human vitreous; vitreomacular adhesion; vitreoretinal contact; vitreoretinal interface; hyalocytes; collagen
MeSH Terms: interventions — Microscopy, Electron, Scanning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cadaver eyes (Experimental): The Central region of the retina and preretinal structures of cadaver eyes are examined
  Interventions: Other: scanning electron microscopy

INTERVENTIONS:
Other: scanning electron microscopy — scanning electron microscopy of the сentral retina and preretinal structures

SUMMARY:
Investigation of the vitreoretinal contact microarchitecture in the macular and paramacular zones of the human retina.

DETAILED DESCRIPTION:
Purpose: to study the features of the macular ILM, to study the features of the preretinal structures of the vitreous body of the Central retinal region, morphofunctional features of preretinal hyalocytes, and the mechanism of vitreoretinal adhesion.

Study Protocol: examination of donor human eyes obtained from an eye Bank after sampling material for corneal transplantation.

Research method: scanning electron microscopy (SEM) of the central retina (macular and paramacular zone): ILM, preretinal vitreous.

Scientific hypothesis: vitreoretinal adhesion is provided not by laminin and fibronectin, but by the interweaving of vitreous collagen fibers between the epiretinal vitreous (more firmly fixed to the retinal surface) and the cortical vitreous.

Expected results: determination of ILM thickness in the macular zone, microanatomy of preretinal vitreous strutcures, and possible mechanism of vitreoretinal adhesion, establishing the possibility of intravital synthesis of collagen fibers synthesis in the adult vitreous.

ELIGIBILITY:
Inclusion Criteria:

* eyes from donors without concomitant multiple organ pathology and ophthalmic pathology

Exclusion Criteria:

* eye injury, age over 45 years, concomitant multiple organ pathology, previous eye diseases

Ages: 35 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
the ILM thickness in the macular zone (foveola) | within 3 days after receiving the cadaver eyes
  the ILM thickness in the macular zone (foveola) in mkm by scanning electron microscopy data
superficial microstructure of ILM | within 3 days after receiving the cadaver eyes
  by scanning electron microscopy data
features of the structural microarchitecture of the preretinal vitreous in the macular zone | within 3 days after receiving the cadaver eyes
  by scanning electron microscopy data
morphofunctional features of preretinal hyalocytes. | within 3 days after receiving the cadaver eyes
  by scanning electron microscopy data

CONTACTS AND LOCATIONS:
Overall Officials: Pavel V Lyskin, PhD, Principal Investigator — The S.N. Fyodorov Eye Microsurgery State Institution
Locations (1):
- S.N. Fedorov Nmrc "Mntk "Eye Microsurgery", Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Microanatomy of vitreoretinal interactions in macular and paramacular areas (article DOI: 10.17816/KMJ2019-595) — https://kazanmedjournal.ru/kazanmedj/article/viewFile/15523/12127
- See also: Microanatomy of Internal Limiting Membrane (article) — https://doi.org/10.25276/0235-4160-2019-1-39-43
- See also: Cellular Microanatomy of Vitreoretinal Interface. Morphofunctional Identification of Epiretinal Vitreous Cells. Collagen Synthesis in Adult Human Vitreous (article) — https://doi.org/10.25276/2307-6658-2019-2-52-56
- See also: New Data of Mechanism in Vitreoretinal Adhesion and Posterior Vitreous Detachment in Humans (article) — https://doi.org/10.25276/2307-6658-2019-2-57-62
- See also: Antithesis to the thesis about fibronectin and laminin as the main components providing vitreoretinal adhesion (article) — https://doi.org/10.25276/2307-6658-2018-4-27-32